CLINICAL TRIAL: NCT00596180
Title: Hyperbaric Oxygen Therapy and SPECT Brain Imaging in Carbon Monoxide Poisoning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paul G. Harch, M.D. (Other)
Collaborators: Harch Hyperbaric Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Other Study IDs: LSU IRB #6626
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Neuropsychiatric Sequelae of Carbon Monoxide Poisoning
Keywords: carbon monoxide poisoning; brain injury
MeSH Terms: conditions — Carbon Monoxide Poisoning; Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: HBOT
  Interventions: Drug: HBOT

INTERVENTIONS:
Drug: HBOT — total body exposure to greater than atmospheric pressure oxygen

SUMMARY:
That SPECT brain imaging tracks and is consistent with clinical history and physical exam as well as cognitive testing.

DETAILED DESCRIPTION:
The study is a retrospective review of the PI's experience using SPECT brain imaging and hyperbaric oxygen therapy in the diagnosis and treatment of non-acute phases of carbon monoxide poisoning. The purpose is to see if the SPECT brain imaging is consistent with the clinical condition and cognitive testing on the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with non-acute carbon monoxide poisoning who underwent SPECT brain imaging as part of their evaluation and treatment

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with non-acute carbon monoxide poisoning who underwent SPECT brain imaging as part of their evaluation and treatment. Retrospective chart review
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
SPECT brain imaging | after completion of HBOT

SECONDARY OUTCOMES:
clinical history and physical exam | after completion of HBOT
Neuropsychological testing | After the final HBOT
  Neuropsychological testing performed after the final HBOT in those who had neuropsychological testing before HBOT

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, M.D., Principal Investigator — LSU School of Medicine
Locations (1):
- Family Physicians Center, Marrero, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No